CLINICAL TRIAL: NCT06536790
Title: Comparative Effects of Hang Clean and Half Squat Training Program on Vertical Jump Performance and Strength Among Basketball Players
Brief Title: Comparative Effects of Hang Clean and Half Squat Training Program Among Basketball Players
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR & AHS/23/0474
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Weight-Bearing Strengthening Program; Muscle Strength; Basketball
Keywords: Weight lifting; Resistance training; Basketball players

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: the assessor who will take the readings is blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hang clean training (Experimental): Group A will perform hang clean training. Three sessions per week for twelve weeks.
  Interventions: Other: hang clean training
- Half squat training (Experimental): Group B will perform half squat training. Three sessions per week for twelve weeks.
  Interventions: Other: half squat training

INTERVENTIONS:
Other: hang clean training — This include hang clean training thrice a week for twelve weeks
  Arms: Hang clean training
Other: half squat training — This include half squat training thrice a week for twelve weeks
  Arms: Half squat training

SUMMARY:
The goal of this randomized controlled trial is to compare the effects of hang clean and half squat training programs on vertical jump performance and strength in male basketball players aged 18-35 years. The main questions it aims to answer are: Does a hang clean training program improve vertical jump performance in basketball players? Does a half squat training program improve vertical jump performance in basketball players? Researchers will compare the hang clean training group to the half squat training group to see if there is a significant difference in the improvement of vertical jump performance and strength. Participants who meet the inclusion criteria will be enrolled and allocated in group A & B through sealed envelop method by Non-probability Convenient random sampling technique. Subjects in Group A will receive hang clean training. Group B will receive half squat training, attend pre- and post-testing assessments of vertical jump performance and strength

DETAILED DESCRIPTION:
Explosive strength is a crucial factor in basketball performance, and various training programs have been developed to improve it. The goal of this randomized controlled trial is to determine the effectiveness of a 12-weeks hang clean training program versus a 12-week half squat training program in improving vertical jump performance and strength in male basketball players aged 18-35 years. The main questions it aims to answer are: Is hang clean training effective in improving vertical jump performance and strength in basketball players? Is half squat training effective in improving vertical jump performance and strength in basketball players? Researchers will compare the hang clean training group to the half squat training group to see if there is a significant difference in the improvement of vertical jump performance and strength. Ethical approval is taken from ethical committee of Riphah International University, Lahore. Participants who meet the inclusion criteria will be enrolled and allocated in group A & B through sealed envelop method by Non-probability Convenient random sampling technique. Study will be carried in basketball courts at Lahore. Participants will be randomly assigned to either the HCL or HSQ training group. Group A will receive hang clean training. Group B will receive half squat training.

ELIGIBILITY:
Inclusion Criteria:

* Male Basketball player
* Having experience with Weight-lifting movements, Squats, and Deadlifts
* No history of anterior cruciate ligament injuries
* No present complaint of Injury.
* 3 years of Professional experience
* Current competitive level

Exclusion Criteria:

* Medical condition
* Previous history of LBP
* Orthopedic or health related conditions
* Female
* Inadequate Training Experience
* Exclude Performance-Enhancing Substance

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2024-09-14 (Estimated); Study Completion 2024-09-14 (Estimated)

PRIMARY OUTCOMES:
vertical jump test | 0 week, 12week
  The vertical jump and reach test through wall will be used to assess the maximum vertical jump height of each participant. The test will be performed by having participants stand side on to a wall with their feet shoulder-width apart. They will reach up with one hand and mark the highest point they can reach with their fingers on the wall. Then, they will perform a maximum vertical jump, landing on both feet, and mark the highest point they can reach at the peak of their jump on the wall. The difference between the two marks will be recorded as the vertical jump height in centimeters (cm). This metric will be used to quantify the improvement in vertical jump performance following the 12-week hang clean training program versus the 12-week half squat training program.
1-repitition maximum for strength | 0 week, 12week
  The 1RM strength metric will be used to quantify the maximum weight an individual can lift in a single repetition of a specific exercise, in this case, the hang clean and half squat exercises. This metric will be used to assess the improvement in maximum strength following the 12-week hang clean training program versus the 12-week half squat training program.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Hamza Afzal, DPT, Principal Investigator — Riphah International University
Locations (1):
- Don Bosco Basketball Court, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ciacci S, Bartolomei S. The effects of two different explosive strength training programs on vertical jump performance in basketball. J Sports Med Phys Fitness. 2018 Oct;58(10):1375-1382. doi: 10.23736/S0022-4707.17.07316-9. Epub 2017 Jun 8. PMID 28597614
- [Background] Perez-Castilla A, Garcia-Ramos A, Padial P, Morales-Artacho AJ, Feriche B. Load-Velocity Relationship in Variations of the Half-Squat Exercise: Influence of Execution Technique. J Strength Cond Res. 2020 Apr;34(4):1024-1031. doi: 10.1519/JSC.0000000000002072. PMID 28885389
- [Background] Hayashi R, Yoshida T, Kariyama Y. Differences in Kinetics during One- and Two-Leg Hang Power Clean. Sports (Basel). 2021 Mar 27;9(4):45. doi: 10.3390/sports9040045. PMID 33801591
- [Background] Petway AJ, Freitas TT, Calleja-Gonzalez J, Medina Leal D, Alcaraz PE. Training load and match-play demands in basketball based on competition level: A systematic review. PLoS One. 2020 Mar 5;15(3):e0229212. doi: 10.1371/journal.pone.0229212. eCollection 2020. PMID 32134965
- [Background] Philipp NM, Cabarkapa D, Nijem RM, Blackburn SD, Fry AC. Vertical Jump Neuromuscular Performance Characteristics Determining On-Court Contribution in Male and Female NCAA Division 1 Basketball Players. Sports (Basel). 2023 Dec 4;11(12):239. doi: 10.3390/sports11120239. PMID 38133106
- [Background] Cabarkapa D, Eserhaut DA, Fry AC, Cabarkapa DV, Philipp NM, Whiting SM, Downey GG. Relationship between Upper and Lower Body Strength and Basketball Shooting Performance. Sports (Basel). 2022 Sep 20;10(10):139. doi: 10.3390/sports10100139. PMID 36287752
- [Background] Stojanovic E, Stojiljkovic N, Scanlan AT, Dalbo VJ, Berkelmans DM, Milanovic Z. The Activity Demands and Physiological Responses Encountered During Basketball Match-Play: A Systematic Review. Sports Med. 2018 Jan;48(1):111-135. doi: 10.1007/s40279-017-0794-z. PMID 29039018
- [Background] Ferioli D, Bosio A, Bilsborough JC, La Torre A, Tornaghi M, Rampinini E. The Preparation Period in Basketball: Training Load and Neuromuscular Adaptations. Int J Sports Physiol Perform. 2018 Sep 1;13(8):991-999. doi: 10.1123/ijspp.2017-0434. Epub 2018 Sep 10. PMID 29345555
- [Background] Barrera-Dominguez FJ, Almagro BJ, Saez de Villarreal E, Molina-Lopez J. Effect of individualised strength and plyometric training on the physical performance of basketball players. Eur J Sport Sci. 2023 Dec;23(12):2379-2388. doi: 10.1080/17461391.2023.2238690. Epub 2023 Jul 30. PMID 37470434
- [Background] Takeuchi K, Tsukuda F. Comparison of the effects of static stretching on range of motion and jump height between quadriceps, hamstrings and triceps surae in collegiate basketball players. BMJ Open Sport Exerc Med. 2019 Dec 22;5(1):e000631. doi: 10.1136/bmjsem-2019-000631. eCollection 2019. PMID 31908836
- [Background] Brini S, Boullosa D, Calleja-Gonzalez J, Ramirez-Campillo R, Nobari H, Castagna C, Clemente FM, Ardigo LP. Neuromuscular and balance adaptations following basketball-specific training programs based on combined drop jump and multidirectional repeated sprint versus multidirectional plyometric training. PLoS One. 2023 Mar 15;18(3):e0283026. doi: 10.1371/journal.pone.0283026. eCollection 2023. PMID 36921008